CLINICAL TRIAL: NCT05091892
Title: The Effect of a Specific Hydrotherapy Program on the Movement From Lying Down to Sitting Position for Children With Cerebral Palsy
Brief Title: Hydrotherapy CP and Lying Down to Sitting Position
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Konstantinos Chandolias, Dr Konstantinos Chandolias, University of Thessaly
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: KC140180
Record Dates: First submitted 2021-10-21; First posted 2021-10-25 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Cerebral Palsy
Keywords: Cerebral palsy; hydrotherapy; Neurodevelopmental treatment; Lying down; Sitting
MeSH Terms: conditions — Cerebral Palsy; Pressure Ulcer

STUDY DESIGN:
Intervention Model Description: 2 equal groups
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Water Group (Experimental): Neurodevelopmental treatment
  Interventions: Other: Hydrotherapy programm
- Land Group (Experimental): Lonqitudinal, transversal and compined rotation in a hydrotherapy programm
  Interventions: Other: Hydrotherapy programm

INTERVENTIONS:
Other: Hydrotherapy programm — Treatment
  Other Names: Neurodevelomental treatment

SUMMARY:
The purpose of this study is to investigate the effect of a very specific hydrotherapy programm on the movement from lying down to sitting position for children with CP

DETAILED DESCRIPTION:
40 children aged 5-11 years with cerebral palsy and difficulty in the transfer activity from lying down to sitting position were randomly divided into 2 groups of 20 children, a land group and a water group. The children of the land attended a neurodevelopmental treatment program and the water group a very specific program in hydrotherapy on combined rotation at all levels. The water program was implemented by specialized physiotherapists in hydrotherapy. The duration of the program for both groups was 3 months. On the first and last day of the intervention, an evaluation of all children was performed using the GMFM and PBS evaluation tests of the evaluation parameters of the transfer from the lying position to the sitting position.

ELIGIBILITY:
Inclusion Criteria:

* Cerebral palsy
* DIfficulties from lying down to sitting posistion

Exclusion Criteria:

* Surgery or injection of botilium toxin in the last year.
* Scheduled surgery or injection of botilium toxin.
* Uncontrolled seizures.
* Do not run elementary commands or play a test representation.
* Autism.
* Syndromes without OP.
* Serious vision problem.
* Absence from the treatment program for more than a week.

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
GMFM | 3 months
  Gross Motor Function Measurement
PBS | 3 months
  Paediatric Balance test

CONTACTS AND LOCATIONS:
Locations (1):
- Konstantinos Chandolias, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: Undecided